CLINICAL TRIAL: NCT02667782
Title: Use of a Mindfulness-based Intervention for Family Carers of People With Dementia in the Community: A Feasibility Study
Brief Title: Feasibility Study on the Use of Mindfulness-based Intervention for Family Carers of People With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Griffith University (Other)
Responsible Party: Principal Investigator, Wai-Tong Chien, Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1-ZVG9
Record Dates: First submitted 2016-01-21; First posted 2016-01-29 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Anxiety; Depression; Dependency Burden; Stress, Psychological
Keywords: Mindfulness-based interventions; Dementia; Caregiving; Burden; Stress; Anxiety; Depression; Community care
MeSH Terms: conditions — Anxiety Disorders; Depression; Stress, Psychological; Dementia | interventions — Mindfulness-Based Stress Reduction; Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-Based Stress Reduction (Experimental): Mindfulness-Based Stress Reduction (MBSR) is developed by Jon Kabat-Zinn in 1979 (Kabat-Zinn, 1990). It is an eight-week Program that includes practices such as gentle mindful movement (awareness of the body), a body scan (to systematically nurture awareness of the body region by region), and sitting meditation (awareness of the breath to include the four foundations of mindfulness, namely, body, feeling tone, mental state, and mental content) (Cullen, 2011).
  Interventions: Behavioral: Mindfulness-Based Stress Reduction (MBSR)
- Mindfulness-Based Cognitive Therapy (Experimental): Mindfulness-Based Cognitive Therapy (MBCT), developed by Zindel Segal, Mark Williams and John Teasdale, employs a cognitive theoretical framework (Cullen, 2011; Segal, Williams, & Teasdale, 2002). It is also delivered as an eight-session group treatment. The first four sessions teach the fundamental concepts and skills of the practice of mindfulness. The remaining four sessions teach the individual how to notice his/her own thoughts and the impact of such thoughts on his/her own physical and emotional experiences.
  Interventions: Behavioral: Mindfulness-Based Cognitive Therapy (MBCT)

INTERVENTIONS:
Behavioral: Mindfulness-Based Stress Reduction (MBSR) — Recruited subjects that are randomly allocated into the MBSR group will have an intensive face-to-face (F-T-F) teaching-learning program that is focused on stress reduction. After that, there will be some regular telephone follow-ups for a closed group of 10-15 participants. Subjects would receive four consecutive weekly F-T-F sessions, then a weekly telephone follow-up for three months in combination with an F-T-F session once a month. The Interventionist will be an experienced mindfulness therapist who is qualified to deliver both MBSR and MBCT.
  Arms: Mindfulness-Based Stress Reduction
Behavioral: Mindfulness-Based Cognitive Therapy (MBCT) — Recruited subjects that are randomly allocated into the MBCT group will have an intensive face-to-face (F-T-F) teaching-learning program that is focused on cognitive therapy. After that, there will be some regular telephone follow-ups for a closed group of 10-15 participants. Subjects would receive four consecutive weekly F-T-F sessions, then a weekly telephone follow-up for three months in combination with an F-T-F session once a month. The Interventionist will be an experienced mindfulness therapist who is qualified to deliver both MBSR and MBCT.
  Arms: Mindfulness-Based Cognitive Therapy

SUMMARY:
The aim of this study is to examine which mindfulness-based intervention protocol, MBCT or MBSR, is more suited for use among local carers of people with dementia (PWD), as measured by better mental health outcomes in PWD such as reductions in stress and improvements in mental well-being.

DETAILED DESCRIPTION:
60 subjects will be recruited in the community and randomized into either the MBCT or MBSR group. Both MBSR and MBCT will be delivered through a face-to-face teaching session followed by regular telephone follow-ups.

The primary outcome measures of the dementia caregivers will be stress with Perceived Stress Scale (PSS; Cohen & Williamson, 1988). The secondary outcome measures of the dementia caregiver will be 1) anxiety with Hospital Anxiety and Depression Scale (HADS; Zigmon & Snaith, 1983), 2) depression with Center for Epidemiologic Studies Depression Scale (CESD; Radloff, 1977), and 3) burden with Zarit Burden Inventory (ZBI; Zarit, Reever, & Bach-Peterson, 1980). The control measure will be their level of mastery of the five facets mindfulness with Five Facets Mindfulness Questionnaire (FFMQ; Baer, Smith, Hopkins, Krietemeyer, & Toney, 2006). Focus group interviews with each group of participants will be conducted post-intervention to explore their experiences and perceptions.

Data will be collected at baseline (T0), at 2 months (the mid-point of the intervention; T1), 4 months (immediately after the intervention; T2), and 7 months (the follow-up assessment; T3). Adherence rates, response rates, and drop-out rates will be collected and analyzed. The triangulation of both qualitative and quantitative data will be performed to determine the suitability and benefits of MBSR and MBCT for carers of PWD in the local setting.

ELIGIBILITY:
one participant (family carer) for each PWD (dementia of any type) living in the community

Inclusion Criteria for the family carer:

* is the primary carer
* of an adult with a confirmed diagnosis of dementia.

Exclusion Criteria:

* has a major active psychiatric illness such as bipolar disorder or schizophrenia.
* is currently undergoing cancer treatment.
* has severe chronic pain (lasting more than six months).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2016-02-18 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Change of Perceived Stress Scale (PSS) | [Time Frame: At baseline (T0), 2 months (mid-point of intervention; T1), 4 months (immediately post- intervention; T2), and 7 months (follow-up assessment; T3).
  Comparisons of changes of Perceived Stress Scale will be considered as follows:
  1. T0 - T1
  2. T0 - T2
  3. T0 - T3
  4. T1 - T2
  5. T1 - T3
  6. T2 - T3

SECONDARY OUTCOMES:
Change of Hospital Anxiety and Depression Scale (HADS) | At baseline (T0), 2 months (mid-point of intervention; T1), 4 months (immediately post- intervention; T2), and 7 months (follow-up assessment; T3).
  Comparisons of changes of Hospital Anxiety and Depression Scale will be considered as follows:
  1. T0 - T1
  2. T0 - T2
  3. T0 - T3
  4. T1 - T2
  5. T1 - T3
  6. T2 - T3
Center for Epidemiologic Studies Depression Scale (CESD) | At baseline (T0), 2 months (mid-point of intervention; T1), 4 months (immediately post- intervention; T2), and 7 months (follow-up assessment; T3).
  Comparisons of changes of Center for Epidemiologic Studies Depression Scale will be considered as follows:
  1. T0 - T1
  2. T0 - T2
  3. T0 - T3
  4. T1 - T2
  5. T1 - T3
  6. T2 - T3
Zarit Burden Inventory (ZBI) | At baseline (T0), 2 months (mid-point of intervention; T1), 4 months (immediately post- intervention; T2), and 7 months (follow-up assessment; T3).
  Comparisons of changes of Zarit Burden Inventory will be considered as follows:
  1. T0 - T1
  2. T0 - T2
  3. T0 - T3
  4. T1 - T2
  5. T1 - T3
  6. T2 - T3

CONTACTS AND LOCATIONS:
Overall Officials: Wai Tong Chien, PhD, Principal Investigator — School of Nursing, The Hong Kong Polytechnic University; Wendy Moyle, PhD, Principal Investigator — Griffith University; Daphne Cheung, PhD, Principal Investigator — School of Nursing, The Hong Kong Polytechnic University
Locations (2):
- Hong Kong (2):
  - School of Nursing, The Hong Kong Polytechnic University, Hong Kong
  - Community care centres, Kowloon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cullen M. (2011). Mindfulness- Based Interventions: an Emerging Phenomenon. Mindfulness. 2(3):186-93.
- [Background] Cohen, S. and Williamson, G. Perceived Stress in a Probability Sample of the United States. Spacapan, S. and Oskamp, S. (Eds.) The Social Psychology of Health. Newbury Park, CA: Sage, 1988
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Radloff, L. S. (1977). The CES-D scale: A self report depression scale for research in the general population. Applied Psychological Measurements, 1, 385-401.
- [Background] Zarit SH, Reever KE, Bach-Peterson J. Relatives of the impaired elderly: correlates of feelings of burden. Gerontologist. 1980 Dec;20(6):649-55. doi: 10.1093/geront/20.6.649. No abstract available. PMID 7203086
- [Background] Baer RA, Smith GT, Hopkins J, Krietemeyer J, Toney L. Using self-report assessment methods to explore facets of mindfulness. Assessment. 2006 Mar;13(1):27-45. doi: 10.1177/1073191105283504. PMID 16443717
- [Background] Segal Z. V., Williams J. M. G., & Teasdale J. D. (2002). Mindfulness-based cognitive therapy for depression: A new approach to preventing relapse. New York: Guilford.
- [Background] Kabat-Zinn, J. (1990). Full Catastrophe Living: How to Cope with Stress, Pain and Illness Using Mindfulness Meditation. New York, NY: Delacorte.